CLINICAL TRIAL: NCT00080119
Title: A Randomized, Double Blind, Placebo Controlled Trial to Determine the Efficacy of Isoniazid (INH) in Preventing Tuberculosis Disease and Latent Tuberculosis Infection Among Infants With Perinatal Exposure to HIV
Brief Title: Daily Isoniazid to Prevent Tuberculosis in Infants Born to Mothers With HIV
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Data Safety Monitoring Board (DSMB) recommended stopping study due to futility
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Comprehensive International Program of Research on AIDS (Other); Secure the Future Foundation (Other)
Responsible Party: Wende Levy, IMPAACT
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PACTG P1041; U01AI068632 (NIH)
Record Dates: First submitted 2004-03-23; First posted 2004-03-25 (Estimated); Results first posted 2010-10-19 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: HIV Infection; Tuberculosis; Pneumocystis Jiroveci Pneumonia
Keywords: Treatment Naive; INH Prophylaxis; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Tuberculosis; Pneumonia, Pneumocystis | interventions — Isoniazid; Trimethoprim; Sulfamethoxazole; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HIVneg/INH (Experimental): Perinatally exposed, HIV-uninfected (HIVneg) children receiving Isoniazid (INH)10-20 mg/kg orally once a day for 96 weeks + Trimethoprim/Sulfamethoxazole (TMP/SMX) 5 mg/kg of TMP component orally once a day until HIV status is confirmed and child is no longer at risk of acquiring HIV through breastfeeding
  Interventions: Drug: Isoniazid (INH); Drug: Trimethoprim/Sulfamethoxazole (TMP/SMX)
- HIVneg/PL (Placebo Comparator): Perinatally exposed, HIV-uninfected (HIVneg) children receiving Isoniazid placebo (PL) orally once a day for 96 weeks + TMP/SMX 5 mg/kg of TMP component orally once a day until HIV status is confirmed and child is no longer at risk of acquiring HIV through breastfeeding
  Interventions: Drug: Isoniazid Placebo (PL)
- HIVpos/INH (Experimental): HIV-infected (HIVpos) children receiving Isoniazid (INH) 10-20 mg/kg orally once a day for 96 weeks + TMP/SMX 5 mg/kg of TMP component orally once a day until one year of age. TMP/SMX may have been continued after one year of age according to WHO guidelines.
  Interventions: Drug: Isoniazid (INH); Drug: Trimethoprim/Sulfamethoxazole (TMP/SMX)
- HIVpos/PL (Placebo Comparator): HIV-infected (HIVpos) children receiving Isoniazid placebo (PL) orally once a day for 96 weeks + TMP/SMX 5 mg/kg of TMP component orally once a day until one year of age. TMP/SMX may have been continued after one year of age according to WHO guidelines.
  Interventions: Drug: Isoniazid Placebo (PL)

INTERVENTIONS:
Drug: Isoniazid (INH) — Antibiotic for the prevention and treatment of TB
  Arms: HIVneg/INH; HIVpos/INH
Drug: Trimethoprim/Sulfamethoxazole (TMP/SMX) — Antibiotic for the prevention and treatment of pneumocystis pneumonia (PCP)
  Arms: HIVneg/INH; HIVpos/INH
Drug: Isoniazid Placebo (PL) — Isoniazid placebo and TMP/SMX
  Arms: HIVneg/PL; HIVpos/PL

SUMMARY:
Tuberculosis (TB) is highly endemic in sub-Saharan Africa. The increased burden of TB in settings with high prevalence of the Human Immunodeficiency Virus (HIV) is associated with high rates of transmission of Mycobacterium tuberculosis (M.tb) to both adults and children. Children infected with TB have a higher risk of developing severe disease than adults with TB. The purpose of this study was to determine if the antibiotic isoniazid (INH) prevented TB infection in infants born to HIV-infected mothers.

DETAILED DESCRIPTION:
Tuberculosis (TB) and the Human Immunodeficiency Virus (HIV) are major public health problems in southern Africa, and the incidence of TB in South Africa is among the highest in the world. TB is caused by the highly contagious bacterium Mycobacterium tuberculosis. The use of Isoniazid (INH) prophylaxis in adults has been associated with reduced risk of TB disease in high-risk populations. Delay in initiating INH prophylaxis in children has resulted in more cases of childhood TB infection. This study evaluated the effectiveness of INH prophylaxis in preventing TB infection in infants born to HIV-infected mothers in southern Africa.

Infants were randomly assigned to receive either INH or placebo by mouth daily, beginning between the 91st and 120th day of life, and at least 90 days after Bacille Calmette-Guerin (BCG) vaccination. At sites in South Africa, HIV-infected infants received daily trimethoprim/sulfamethoxazole (TMP/SMX) as Pneumocystis jiroveci pneumonia (PCP) prophylaxis until at least 1 year of age; HIV-uninfected infants received TMP/SMX until at least 6 months of age.

The study was to follow participants for 192 weeks. Study visits occurred at study entry and every 12 weeks until week 192. A physical exam and blood collection occurred at each study visit. Infants were assessed for peripheral neuropathy every 12 weeks until week 96 and for TB at weeks 96, 144, and 192. The study also assessed medication adherence.

As of November 12, 2008, follow-up was revised. All participants were permanently discontinued from study follow-up by February 28, 2009 and no later than May 31, 2009. Only clinical evaluations were performed for all participants. For HIV-infected participants, the study drug was stopped at the next scheduled visit. For HIV-uninfected subjects, the study drug was discontinued immediately.

ELIGIBILITY:
Inclusion Criteria:

* Mother is HIV-infected. Hard copy documentation of the mother's HIV infection is unnecessary if a positive DNA PCR from her infant is available.
* Received Bacille Calmette-Guerin (BCG) vaccine up to and including the 30th day of life and at least 90 days prior to study entry
* Able to complete all study requirements
* Physician assessment of age-appropriate neurodevelopment in which the chronological age is corrected for gestational age for prematurely born infants
* Parent or legal guardian able and willing to provide signed informed consent
* Plan to live in the study area for at least 4 years
* For inclusion in HIV-infected stratum, infant must have a positive HIV-1 DNA PCR; for inclusion in HIV-uninfected stratum, infant must have a negative HIV-1 DNA PCR performed at >= 4 weeks of age

Exclusion Criteria:

* Previous diagnosis of TB infection, TB disease or current treatment for TB infection or TB disease
* Previous receipt of INH
* Contact with a known acid fast bacilli (AFB) sputum smear or culture-positive case of TB before study entry
* Current acute or recurrent (3 or more prior episodes) lower respiratory tract disease
* Chronic persistent diarrhea
* Failure to thrive
* Contraindications for use of INH or TMP/SMX
* Require certain medications
* Known or suspected immune system diseases other than HIV
* Current or previous diagnosis of or treatment for cancer
* Current immunosuppressive therapy greater than 1 mg/kg/day of prednisone or equivalent
* Anticipated long-term oral or intravenous corticosteroid therapy (greater than 3 weeks). Those receiving nonsteroidal anti-inflammatory agents and inhaled corticosteroids are not excluded.
* Grade 3 or greater AST/SGOT, ALT/SGPT, ANC, hemoglobin, platelet count, rash, neuropathy, or myopathy at screening
* Any Grade 4 clinical or laboratory toxicity within 14 days prior to study entry
* Other acute or chronic conditions that, in the opinion of the investigator, may interfere with the study

Ages: 91 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1354 (Actual)
Dates: Start 2004-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shabir Madhi, MD, Study Chair — University of Witwatersrand, South Africa; George McSherry, MD, Study Chair — UMDNJ - New Jersey Medical School; Charles D. Mitchell, MD, Study Chair — University of Miami
Locations (6):
- Princess Marina Hospital, Gaborone, Botswana
- South Africa (5):
  - University of Cape Town, Red Cross Children's Hospital, Cape Town
  - University of Stellenbosch, Tygerberg Hospital, Cape Town
  - Nelson R. Mandela School of Medicine, University of KwaZulu Natal, Durban, Durban
  - Perinatal HIV Research Unit at Chris Hani Baragwanath Hospital, Johannesburg
  - Chris Hani Baragwanath Hospital, Harriet Shezi Clinic, Johannesburg

REFERENCES:
- [Background] Chintu C, Mwaba P. Tuberculosis in children with human immunodeficiency virus infection. Int J Tuberc Lung Dis. 2005 May;9(5):477-84. PMID 15875917
- [Background] Corbett EL, Watt CJ, Walker N, Maher D, Williams BG, Raviglione MC, Dye C. The growing burden of tuberculosis: global trends and interactions with the HIV epidemic. Arch Intern Med. 2003 May 12;163(9):1009-21. doi: 10.1001/archinte.163.9.1009. PMID 12742798
- [Background] de Jong BC, Israelski DM, Corbett EL, Small PM. Clinical management of tuberculosis in the context of HIV infection. Annu Rev Med. 2004;55:283-301. doi: 10.1146/annurev.med.55.091902.103753. PMID 14746522
- [Background] Toossi Z. Virological and immunological impact of tuberculosis on human immunodeficiency virus type 1 disease. J Infect Dis. 2003 Oct 15;188(8):1146-55. doi: 10.1086/378676. Epub 2003 Sep 30. PMID 14551885
- [Result] Cotton MF, Schaaf HS, Lottering G, Weber HL, Coetzee J, Nachman S; PACTG 1041 Team. Tuberculosis exposure in HIV-exposed infants in a high-prevalence setting. Int J Tuberc Lung Dis. 2008 Feb;12(2):225-7. PMID 18230259
- [Result] Cotton M, Kim S, Rabie H, Coetzee J, Nachman S. A window into a public program for prevention of mother to child transmission of HIV: evidence from a prospective clinical trial. South Afr J HIV Med. 2009 Jan 1;10(4):16-19. doi: 10.4102/sajhivmed.v10i4.257. PMID 20607114
- [Derived] Gupta A, Montepiedra G, Gupte A, Zeldow B, Jubulis J, Detrick B, Violari A, Madhi S, Bobat R, Cotton M, Mitchell C, Spector S; IMPAACT NWCS113 and P1041 Study Team. Low Vitamin-D Levels Combined with PKP3-SIGIRR-TMEM16J Host Variants Is Associated with Tuberculosis and Death in HIV-Infected and -Exposed Infants. PLoS One. 2016 Feb 12;11(2):e0148649. doi: 10.1371/journal.pone.0148649. eCollection 2016. PMID 26872154
- [Derived] Madhi SA, Nachman S, Violari A, Kim S, Cotton MF, Bobat R, Jean-Philippe P, McSherry G, Mitchell C; P1041 Study Team. Primary isoniazid prophylaxis against tuberculosis in HIV-exposed children. N Engl J Med. 2011 Jul 7;365(1):21-31. doi: 10.1056/NEJMoa1011214. PMID 21732834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at four study sites, three in South Africa and one in Botswana, between December 13, 2004 and June 26, 2008
Pre-assignment Details: Infants perinatally exposed to HIV 91-120 days with documented receipt of Bacille Calmette-Guerin (BCG) vaccine by 30 days (>=90 days since receipt), no previous diagnosis or treatment of TB or contact with known TB case, stratified by HIV and randomized to receive blinded INH or INH placebo. 3 participants randomized but did not start treatment.
Groups:
- HIVneg/PL: Perinatally-exposed, HIV-uninfected (HIVneg) children receiving Isoniazid placebo (PL) orally once a day for 96 weeks + TMP/SMX 5 mg/kg of TMP component orally once a day until HIV status is confirmed and child is no longer at risk of acquiring HIV through breastfeeding
Period: Overall Study
Arm/Group | HIVneg/INH | HIVneg/PL | HIVpos/INH | HIVpos/PL
Started | 403 | 401 | 273 | 274
Completed | 347 | 339 | 108 | 111
Not Completed | 56 | 62 | 165 | 163
Not completed — Discontinued because of study closure | 0 | 0 | 130 | 141
Not completed — Unable to get to clinic | 24 | 24 | 7 | 1
Not completed — Consent withdrawn | 13 | 17 | 4 | 6
Not completed — Unwilling to adhere to study requirement | 3 | 2 | 5 | 1
Not completed — Lost to Follow-up | 16 | 19 | 19 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIVneg/INH | HIVneg/PL | HIVpos/INH | HIVpos/PL | Total
Number analyzed (Participants) | 403 | 401 | 273 | 274 | 1351
Age, Customized [Number; unit: participants]
  91-100 days | 258 | 253 | 171 | 192 | 874
  101-110 days | 71 | 84 | 56 | 33 | 244
  111-120 days | 74 | 64 | 46 | 49 | 233
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 190 | 159 | 151 | 703
  Male | 200 | 211 | 114 | 123 | 648
Race/Ethnicity, Customized [Number; unit: participants]
  Indigenous African | 389 | 386 | 264 | 272 | 1311
  Mixed ancestry/other | 14 | 15 | 9 | 2 | 40
Age at receipt of Bacille Calmette-Guerin (BCG) vaccination (days) [Number; unit: participants]
  <= 7 days | 395 | 392 | 255 | 258 | 1300
  8-29 days | 8 | 9 | 18 | 16 | 51
Any smoker in household [Number; unit: participants]
  Yes | 191 | 177 | 120 | 131 | 619
  No | 211 | 224 | 153 | 141 | 729
  Missing | 1 | 0 | 0 | 2 | 3
Birth weight (grams) [Number; unit: participants]
  <2500 grams | 49 | 49 | 68 | 56 | 222
  >= 2500 grams | 354 | 352 | 205 | 218 | 1129
CD4% [Number; unit: participants] — Only for HIV-infected participants. Those in the HIV-infected stratum that were later determined to be HIV-uninfected are recorded as not applicable.
  participants
    <20% | 0 | 0 | 56 | 55 | 111
    20%-<25% | 0 | 0 | 40 | 46 | 86
    >= 25% | 0 | 0 | 162 | 157 | 319
    Missing | 0 | 0 | 14 | 13 | 27
    Not applicable | 403 | 401 | 1 | 3 | 808
Centers for Disease Control (CDC) Disease Category [Number; unit: participants] — Only for HIV-infected participants.
  participants
    Category N or A | 0 | 0 | 252 | 244 | 496
    Category B | 0 | 0 | 16 | 21 | 37
    Category C | 0 | 0 | 2 | 3 | 5
    HIV-uninfected on repeat test | 0 | 0 | 1 | 3 | 4
    Missing | 0 | 0 | 2 | 3 | 5
    Not applicable (HIV-uninfected) | 403 | 401 | 0 | 0 | 804
Caregiver currently smokes [Number; unit: participants]
  Yes | 11 | 25 | 16 | 10 | 62
  No | 392 | 376 | 257 | 264 | 1289
Ever breastfed [Number; unit: participants]
  Yes | 24 | 24 | 37 | 36 | 121
  No | 379 | 377 | 236 | 238 | 1230
HIV-1 RNA (copies/ml) [Number; unit: participants] — Only for HIV-infected participants. Those in the HIV-infected stratum that were later determined to be HIV-uninfected are recorded as not applicable.
  participants
    <= 400 copies/ml | 0 | 0 | 8 | 12 | 20
    401 - <20,000 copies/ml | 0 | 0 | 36 | 51 | 87
    20,000 - < 750,000 copies/ml | 0 | 0 | 91 | 86 | 177
    >= 750,000 copies/ml | 0 | 0 | 129 | 116 | 245
    Missing | 0 | 0 | 8 | 6 | 14
    Not applicable | 403 | 401 | 1 | 3 | 808
History of tuberculosis (TB) in mother [Number; unit: participants]
  Yes | 33 | 25 | 14 | 25 | 97
  No | 370 | 376 | 259 | 249 | 1254
Housing [Number; unit: participants]
  Formal (brick) house | 235 | 233 | 162 | 183 | 813
  Informal (shack/wooden) | 168 | 168 | 109 | 89 | 534
  Hostel | 0 | 0 | 2 | 0 | 2
  Missing | 0 | 0 | 0 | 2 | 2
On antiretrovirals at entry [Number; unit: participants] — Only for HIV-infected participants. Those in the HIV-infected stratum that were later determined to be HIV-uninfected are recorded as not applicable.
  participants
    Yes | 0 | 0 | 78 | 93 | 171
    No | 0 | 0 | 194 | 178 | 372
    Not applicable | 403 | 401 | 1 | 3 | 808
Site of enrollment [Number; unit: participants]
  Johannesburg, S Africa | 259 | 260 | 180 | 179 | 878
  Cape Town, S Africa | 140 | 138 | 66 | 65 | 409
  Durban, S Africa | 4 | 3 | 26 | 27 | 60
  Gaborone, Botswana | 0 | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Development of Tuberculosis (TB) Disease or Death Among HIV-infected Children
Description: Criteria for diagnosis with TB disease: Definite-isolation of Mycobacterium TB (M.tb) or +ve stain on cerebrospinal fluid (CSF); Probable- +ve acid fast bacilli (AFB) stain on fluids/tissues other than CSF and sufficient clinical criteria/radiographic evidence suggestive of TB; Possible-abnormal chest radiograph suggestive of pulmonary TB (PTB) and either a +ve tuberculin skin test (TST) or minimum score on algorithm for clinical TB. Records reviewed by Endpoint Review Group. Results report percent of participants reaching TB disease/death by week 96 calculated using the Kaplan-Meier method.
Time Frame: Through to week 96
Population: Includes HIVpos who started study treatment. Time from randomization to TB disease/death was calculated. Participants lost-to-follow-up (LTF) <96 wks (+12wks) censored at the time of LTF. Participants in follow-up at 96 wks free of TB disease censored at 96 wks. Participants on study when study discontinued censored at discontinuation visit.
Measure: Number; unit: Percent of participants
Arm/Group | HIVpos/INH | HIVpos/PL
Number analyzed (Participants) | 273 | 274
Percent of participants | 27.4 | 28.9
Statistical Analysis 1: Comparison: HIVpos/INH vs HIVpos/PL; Test type: Superiority or Other; p = 0.93, Log Rank — Threshold p-value for significance = 0.0492; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.67 to 1.44] — Hazard ratio for INH relative to Placebo

2. Primary Outcome: Time From Randomization to Development of TB Infection or Death Among Perinatally Exposed, HIV-uninfected Children
Description: Criteria for diagnosis with TB infection were outlined in the protocol. TB infection included TB disease (see primary outcome measure 1 for definition) and latent TB infection. Latent TB infection was diagnosed by a positive tuberculin skin test (TST) based on a purified protein derivative (PPD) performed at week 96. Participant records were reviewed by an Endpoint Review Group to verify that participants had met the criteria for TB infection. Results report percent of participants reaching TB infection or death by week 96 calculated using the Kaplan-Meier method.
Time Frame: Through to week 96
Population: HIVneg who started study treatment were included. Time from randomization to first of TB infection/death was calculated. Participants lost-to-follow-up before 96 wks were censored at the time of loss-to-follow-up. Participants in follow-up at 96 weeks (+12 week window) who were free of TB infection were censored at 96 weeks (+12 week window).
Measure: Number; unit: Percent of participants
Arm/Group | HIVneg/INH | HIVneg/PL
Number analyzed (Participants) | 403 | 401
Percent of participants | 10.9 | 12.6
Statistical Analysis 1: Comparison: HIVneg/INH vs HIVneg/PL; Test type: Superiority or Other; p = 0.43, Log Rank — Threshold p-value for significance = 0.0493; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.55 to 1.30] — Hazard ratio for INH relative to Placebo

3. Secondary Outcome: Time From Randomization to Development of TB Infection or Death Among HIV-infected Children
Description: Criteria for diagnosis with TB infection were outlined in the protocol. TB infection included TB disease (see primary outcome measure 1 for definition) and latent TB infection. Latent TB infection was diagnosed by a positive TST based on a PPD performed at week 96. Participant records were reviewed by an Endpoint Review Group to verify that participants had met the criteria for TB infection. Results report percent of participants reaching TB infection or death by week 96 calculated using the Kaplan-Meier method.
Time Frame: Through to week 96
Population: HIVpos starting study treatment were included. Time from randomization to first of TB infection/death was calculated. Participants LTF <96 weeks (+12 wk) censored at the time LTF. Participants in follow-up at 96 wks free of TB infection censored at 96 wks. Participants on study when study discontinued were censored at discontinuation visit.
Measure: Number; unit: Percent of participants
Arm/Group | HIVpos/INH | HIVpos/PL
Number analyzed (Participants) | 273 | 274
Percent of participants | 29.4 | 32.8

4. Secondary Outcome: Time From Randomization to HIV Disease Progression or Death Among HIV-infected Children
Description: HIV disease progression was defined as any advancement in Centers for Disease Control (CDC) disease category from entry or death. If a participant was CDC disease category C at entry progression was defined as death. Results report percent of participants with HIV progression or death by week 96 calculated using the Kaplan-Meier method.
Time Frame: Through to week 96
Population: Includes HIVpos starting study treatment. Time from randomization to first of disease progression/death calculated. Censored if LTF <96 wks, at 96 wks (if on study) or at discontinuation visit. Participants found to be HIVneg upon repeat testing could only progress by meeting a death endpoint.
Measure: Number; unit: Percent of participants
Arm/Group | HIVpos/INH | HIVpos/PL
Number analyzed (Participants) | 273 | 274
Percent of participants | 30.6 | 22.5

5. Secondary Outcome: Time From Randomization to Development of TB Disease or Death Among Perinatally Exposed, HIV-uninfected Children
Description: Criteria for diagnosis with TB disease were: Definite-isolation of M.tb or positive stain on CSF; Probable-positive AFB stain on fluids/tissues other than CSF and sufficient clinical criteria/radiographic evidence suggestive of TB; Possible-abnormal chest radiograph suggestive of PTB and either a +ve TST or minimum score on algorithm to diagnose clinical TB. All records were reviewed by an Endpoint Review Group to verify that participants had met the criteria for TB disease. Results report percent of participants reaching TB disease/death by week 96 calculated using the Kaplan-Meier method.
Time Frame: Through to week 96
Population: Includes HIVneg who started study treatment. Time from randomization to the first of TB disease/death was calculated. Participants lost-to-follow-up before 96 weeks (+12 week window)were censored at the time of loss-to-follow-up. Participants in follow-up at 96 weeks who were free of TB disease were censored at 96 weeks (+12 week window).
Measure: Number; unit: Percent of participants
Arm/Group | HIVneg/INH | HIVneg/PL
Number analyzed (Participants) | 403 | 401
Percent of participants | 8.3 | 9.1

6. Secondary Outcome: Time From Randomization to Development of TB Disease Among HIV Infected and Perinatally Exposed, HIV-uninfected Children
Description: as for outcome 5
Time Frame: Through to week 96
Population: Includes all starting study treatment. Time from randomization to development of TB disease was calculated. Participants LTF <96 wks (+12 wks) censored at time of LTF. Participants in follow-up at 96 wks free of TB disease censored at 96 wks. HIVpos on study when study discontinued were censored at their discontinuation visit.
Measure: Number; unit: Percent of participants
Arm/Group | HIVneg/INH | HIVneg/PL | HIVpos/INH | HIVpos/PL
Number analyzed (Participants) | 403 | 401 | 273 | 274
Percent of participants | 7.8 | 8.5 | 20.3 | 23.7

7. Secondary Outcome: Time From Randomization to Development of TB Infection Among HIV-infected and Perinatally Exposed, HIV-uninfected Children
Description: Criteria for diagnosis with TB infection were outlined in the protocol. TB infection included TB disease (see primary outcome measure 1 for definition) and latent TB infection. Latent TB infection was diagnosed by a positive TST based on a PPD performed at week 96. Participant records were reviewed by an Endpoint Review Group to verify that participants had met the criteria for TB infection. Results report percent of participants reaching TB infection by week 96 calculated using the Kaplan-Meier method.
Time Frame: Through to week 96
Population: Includes all starting study treatment. Time from randomization to development of TB infection was calculated. Participants LTF <96 weeks (+12 wks) censored at the time of LTF. Participants in follow-up at 96 wks free of TB infection were censored at 96 wks. HIVpos on study when study discontinued censored at their discontinuation visit.
Measure: Number; unit: Percent of participants
Arm/Group | HIVneg/INH | HIVneg/PL | HIVpos/INH | HIVpos/PL
Number analyzed (Participants) | 403 | 401 | 273 | 274
Percent of participants | 10.4 | 12.1 | 22.4 | 27.9

8. Secondary Outcome: Time From Randomization to Death Among HIV-infected and Perinatally Exposed, HIV-uninfected Children
Description: Deaths from any cause were included. Results report percent of participants dying by week 96 calculated using the Kaplan-Meier method.
Time Frame: Through to week 96
Population: Includes all starting study treatment. Time from randomization to death was calculated. Participants LTF <96 weeks (+12 wks) censored at the time of LTF. Participants in follow-up at 96 wks (+12 wks) censored at 96 weeks. HIVpos on study when study was discontinued were censored at their discontinuation visit.
Measure: Number; unit: Percent of participants
Arm/Group | HIVneg/INH | HIVneg/PL | HIVpos/INH | HIVpos/PL
Number analyzed (Participants) | 403 | 401 | 273 | 274
Percent of participants | 0.8 | 0.8 | 11.6 | 7.2

9. Secondary Outcome: Time From Randomization to First New Grade 3 or Worse Adverse Event Among HIV-infected and Perinatally Exposed, HIV-uninfected Children
Description: Signs, symptoms and laboratory values were graded according to the Division of AIDS Adverse Event Grading System. Any event of grade 3 or higher not present at entry that occurred after randomization was classified as a new event. Results report percent of participants with a new event by week 96 calculated using the Kaplan-Meier method.
Time Frame: Through to week 96
Population: Includes all starting treatment. Time from randomization to first new adverse event (AE) calculated. For lab toxicities, censored at visit following permanent discontinuation of study drugs. For signs/symptoms, participants in follow-up at 96 wks (+12) with no new grade >=3 AE censored at 96 wks. Participants LTF <96 wks censored at LTF.
Measure: Number; unit: Percent of participants
Arm/Group | HIVneg/INH | HIVneg/PL | HIVpos/INH | HIVpos/PL
Number analyzed (Participants) | 403 | 401 | 273 | 274
Percent of participants
  New >=grade 3 sign/symptom | 5.0 | 4.2 | 16.8 | 11.7
  New >= grade 3 peripheral neuropathy | 1.1 | 0.3 | 2.4 | 0.8
  New >=grade 3 lab abnormality | 4.9 | 4.6 | 11.3 | 10.1
  New >=grade 3 hemoglobin | 0.0 | 0.0 | 1.8 | 1.2
  New >=grade 3 ANC | 1.7 | 0.3 | 1.6 | 3.5
  New >=grade 3 platelets | 0.3 | 0.0 | 1.7 | 0.9
  New >=grade 3 SGOT | 1.0 | 2.8 | 0.4 | 2.5
  New >=grade 3 SGPT | 2.8 | 4.4 | 5.9 | 4.0

ADVERSE EVENTS:
Time Frame: From study enrollment until study completion and before May 25, 2009 (primary completion date)
Description: Expedited adverse event (AE) reporting followed Intensive Division of AIDS (DAIDS) Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities, requiring hospitalization, and >=grade 3 AEs defined by the "DAIDS Table for Grading the Severity of Adult and Pediatric AEs", V1.0, 12/2004.
Arm/Group | HIVneg/INH | HIVneg/PL | HIVpos/INH | HIVpos/PL
Serious Adverse Events (participants affected / at risk) | 25/403 | 18/401 | 55/273 | 42/274
Other Adverse Events (participants affected / at risk) | 353/403 | 368/401 | 264/273 | 268/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIVneg/INH (N=403) | HIVneg/PL (N=401) | HIVpos/INH (N=273) | HIVpos/PL (N=274)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Accidental death (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 2 | 8 | 6
Sudden infant death syndrome (General disorders) | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 6 | 5 | 6 | 6
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 9 | 6
HIV infection (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 6 | 5
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia herpes viral (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 2 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Tuberculosis of eye (Infections and infestations) | 0 | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 6 | 2 | 2
Transaminases increased (Investigations) | 2 | 1 | 2 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 5 | 1 | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIVneg/INH (N=403) | HIVneg/PL (N=401) | HIVpos/INH (N=273) | HIVpos/PL (N=274)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 10 | 28
Diarrhoea (Gastrointestinal disorders) | 16 | 28 | 18 | 26
AIDS encephalopathy (Infections and infestations) | 0 | 1 | 21 | 24
Acarodermatitis (Infections and infestations) | 22 | 20 | 9 | 15
Bronchiolitis (Infections and infestations) | 40 | 41 | 12 | 12
Bronchitis (Infections and infestations) | 24 | 33 | 18 | 11
Gastroenteritis (Infections and infestations) | 90 | 104 | 81 | 79
Oral candidiasis (Infections and infestations) | 13 | 11 | 54 | 54
Otitis media acute (Infections and infestations) | 140 | 162 | 46 | 53
Pharyngitis (Infections and infestations) | 122 | 131 | 68 | 63
Pneumonia (Infections and infestations) | 11 | 12 | 33 | 28
Pulmonary tuberculosis (Infections and infestations) | 39 | 44 | 47 | 47
Tonsilitis (Infections and infestations) | 99 | 108 | 41 | 41
Upper respiratory tract infection (Infections and infestations) | 26 | 36 | 5 | 4
Alanine aminotransferase increased (Investigations) | 124 | 121 | 130 | 114
Aspartate aminotransferase increased (Investigations) | 88 | 94 | 109 | 86
Gamma-glutamyltransferase increased (Investigations) | 9 | 8 | 14 | 7
Haemoglobin decreased (Investigations) | 70 | 72 | 176 | 176
Neutrophil count decreased (Investigations) | 117 | 100 | 100 | 105
Failure to thrive (Metabolism and nutrition disorders) | 51 | 33 | 41 | 42
Neuropathy peripheral (Nervous system disorders) | 47 | 50 | 75 | 87
Eczema (Skin and subcutaneous tissue disorders) | 41 | 41 | 65 | 49

LIMITATIONS AND CAVEATS:
DSMB recommended stopping study due to futility: "no compelling reason to enroll additional infants" or "to continue to treat participants with the blinded study medication". Week 192 analyses not done as <4% (26%) of HIVpos (HIVneg) reached wk 192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.